CLINICAL TRIAL: NCT00061178
Title: Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Efficacy & Safety of rhuMAb VEGF in Previously Treated Metastatic Renal Cell Carcinoma
Brief Title: Efficacy and Safety Study of rhuMAb VEGF to Treat Metastatic Renal Cell Carcinoma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No patients were enrolled, study cancelled before start
Sponsor: Genentech, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVF2665g
Record Dates: First submitted 2003-05-21; First posted 2003-05-23 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Bevacizumab

INTERVENTIONS:
Drug: rhuMAb VEGF (Bevacizumab)

SUMMARY:
The purpose of this study is to determine whether rhuMAb VEGF (Bevacizumab) is safe and effective for the treatment of renal cell cancer when other treatments have failed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Histologically confirmed, metastatic renal cell cancer (RCC) of clear cell histology
* Clinical or radiographic evidence of disease progression (as assessed by the investigator and reviewed by the Sponsor) during or after completion of one, and only one, cytokine-based regimen for metastatic disease
* At least 21 days since any prior therapy for RCC
* Prior nephrectomy
* Use of an acceptable means of contraception (potentially fertile men and women)
* ECOG performance status of 0 or 1
* Life expectancy >= 3 months
* Age 18 years or older

Exclusion Criteria:

* RCC of papillary or collecting-duct type
* More than one nonsurgical therapy for metastatic RCC (note that medroxyprogesterone acetate not used for physiologic replacement or birth control is considered a therapy for RCC for the purposes of this study)
* Prior treatment with thalidomide
* Radiotherapy within 14 days of Day 0
* Current, recent (within 21 days of Day 0), or planned participation in an experimental drug study
* Pregnant or breast-feeding subjects
* Any of the following screening clinical laboratory values: 24-hour urine collection with >= 1 g of protein; Serum creatinine > 2.0 mg/dL; Absolute neutrophil count (ANC) <500/mL; Platelet count <75,000/mL; INR >= 1.5; Total bilirubin > 2.0 mg/dL; AST or ALT > 5 x the upper limit of normal (ULN) for subjects with documented liver metastases or > 2.5 x the ULN for subjects without evidence of liver metastases; Hemoglobin < 9 gm/dL (may be transfused or receive epoetin alfa [e.g., Epogen] to maintain or exceed this level)
* Other invasive malignancies within 5 years of randomization (other than squamous or basal cell carcinoma of the skin)
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications
* Inability to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)